CLINICAL TRIAL: NCT00146393
Title: Evaluation of People With Arthritis Can Exercise
Brief Title: Health Benefits of an Exercise Program for Adults With Arthritis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: University of North Carolina (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDC-NCCDPHP-0275; CDC-PEP-MM0275
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2005-12-09 (Estimated); Status verified 2005-09

CONDITIONS: Arthritis; Osteoarthritis; Rheumatoid Arthritis
Keywords: exercise; physical activity; physical conditioning; pain; physical function
MeSH Terms: conditions — Arthritis; Osteoarthritis; Arthritis, Rheumatoid; Motor Activity; Pain

INTERVENTIONS:
Behavioral: People with Arthritis Can Exercise program

SUMMARY:
The primary goal of this study is to assess the effect of People with Arthritis Can Exercise (PACE), a community-based group recreational exercise program, on key arthritis-related health outcomes among adults with arthritis.

DETAILED DESCRIPTION:
Self-management is very important in chronic diseases, and promoting physical activity is a key public health strategy for arthritis management. Although several exercise programs such as People with Arthritis Can Exercise (PACE) have been created to implement this strategy, none have sufficient scientific evidence supporting their effectiveness to promote the programs through public health avenues.

The primary goal of this study is to assess the effect of PACE(People with Arthritis Can Exercise), a community-based group recreational exercise program, on key arthritis-related health outcomes. The primary goal of the study will be accomplished through an eight week randomized controlled trial conducted with 480 participants residing in eight urban or rural communities in North Carolina. This project is designed to evaluate the effectiveness of the program in changing arthritis-related health outcomes such as pain, function and physical activity levels. The project will compare the eight week PACE program to a control group.

The specific objectives are as follows: (The aims have not been modified.)

1. To further review the PACE conceptual framework and materials in order to develop a standardized PACE protocol to be delivered in the study as well as to refine study measures.
2. To work closely with the Carolinas AF Chapter to develop collaborative relationships with local health departments and key contacts in communities identified for PACE implementation.
3. To recruit 480 individuals to participate in a randomized controlled trial of PACE in eight communities and to implement the PACE program.
4. To compare changes in key arthritis-related health outcomes between PACE participants and controls over eight weeks (PACE course time frame).
5. To determine longer-term benefits of the PACE intervention by examining key arthritis-related health outcomes 3 and 6 months post completion of the intervention.
6. To conduct qualitative research among PACE completers and non-completers to determine motivators and barriers to success, as well as to determine the acceptability and suitability of the program.
7. To formulate recommendations or modifications for implementation of the PACE program.

ELIGIBILITY:
Inclusion Criteria:

* Adults over age 18
* Have some form of arthritis (examples: osteoarthritis, rheumatoid arthritis, lupus, fibromyalgia, gout, etc.)
* Be able to move independently without assistance
* Currently exercising less than 3 times per week

Exclusion Criteria:

* Inability to walk without assistance
* Severe health condition where exercise is contraindicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347
Dates: Start 2003-07; Study Completion 2004-06

PRIMARY OUTCOMES:
Visual Analog Scale pain level at baseline, 2, 3 and 6 months
Self-reported physical function (Health Assessment Questionnaire) at baseline, and 2, 3 and 6 months
Measured function (6 minute walk, 360 deg turn, walking speed and timed chair stands, 10 lb lift) at baseline and 2 months
Physical activity level (Physical Activity Scale for the Elderly : PASE) at baseline, 2, 3 and 6 months

SECONDARY OUTCOMES:
Visual analog scale fatigue
Visual analog scale stiffness
Rheumatoid Arthritis Self-efficacy Scale (RASE)
Center for Epidemiologic Studies Depression Scale (CES-D)
Outcomes Expectations for Exercise (OEE)
COnfidence Self-efficacy (CSE)
Rheumatology Attitudes Index (RAI)
Tampa Scale for Kinesiophobia (TSK)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M Hootman, PhD, Study Chair — Centers for Disease Control and Prevention; Leigh Callahan, PhD, Principal Investigator — University of North Carolina, Chapel Hill

REFERENCES:
- [Result] Schoster B, Callahan LF, Meier A, Mielenz T, DiMartino L. The People with Arthritis Can Exercise (PACE) program: a qualitative evaluation of participant satisfaction. Prev Chronic Dis. 2005 Jul;2(3):A11. Epub 2005 Jun 15. PMID 15963313
- [Derived] Callahan LF, Mielenz T, Freburger J, Shreffler J, Hootman J, Brady T, Buysse K, Schwartz T. A randomized controlled trial of the people with arthritis can exercise program: symptoms, function, physical activity, and psychosocial outcomes. Arthritis Rheum. 2008 Jan 15;59(1):92-101. doi: 10.1002/art.23239. PMID 18163409